CLINICAL TRIAL: NCT04044625
Title: Effects of High-intensity Versus Low-intensity Noninvasive Positive Pressure Ventilation in Acute Exacerbation of Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial
Brief Title: Effects of High-intensity Noninvasive Positive Pressure Ventilation in AECOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zujin Luo, Principal Investigator, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BeijingCYH-ICU-007
Record Dates: First submitted 2019-05-21; First posted 2019-08-05 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity NPPV (Experimental): The patients will receive high-intensity noninvasive positive pressure ventilation.
  Interventions: Device: High-intensity NPPV
- Low-intensity NPPV (Active Comparator): The patients will receive low-intensity noninvasive positive pressure ventilation.
  Interventions: Device: Low-intensity NPPV

INTERVENTIONS:
Device: High-intensity NPPV — In the high-intensity NPPV group, patients will undergo pressure-limited NPPV (eg, NPPV in spontaneous/timed mode) at a higher IPAP level. IPAP is initially set at 10 cmH2O and continuously adjusted by increments and decrements of 1-2 cmH2O (typically ranging between 20 and 30 cmH2O), according to patients' tolerance, to obtain a tidal volume (VT) of 10-15 mL/kg. IPAP should be increased as much as possible to decrease PaCO2 to a normal level. However, if PaCO2 decreases to less than 35 mmHg, IPAP should be decreased to achieve normocapnia.
  Arms: High-intensity NPPV
Device: Low-intensity NPPV — In the low-intensity NPPV group, patients will undergo pressure-limited NPPV (eg, NPPV in spontaneous/timed mode) with a conventional IPAP level. IPAP is initially set to 10 cmH2O and is continuously adjusted by increments and decrements of 1-2 cmH2O (up to 20 cmH2O), according to patients' tolerance, to obtain a VT of 6-10 mL/kg.
  Arms: Low-intensity NPPV

SUMMARY:
This study aims to investigate the effects of high-intensity noninvasive positive pressure ventilation (NPPV), as compared with low-intensity NPPV, on hypercapnia, consciousness, inspiratory muscle effort, dyspnea, NPPV tolerance, inflammatory response, adverse events and other outcomes in patients with acute exacerbation of chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of COPD according to the criteria of the Global Initiative for Chronic Obstructive Lung Disease in 2019
2. Presence of acute exacerbation
3. Arterial pH <7.35 with arterial carbon dioxide tension (PaCO2) >45 mmHg on room air or supplemental oxygen
4. PaCO2 >45 mmHg following low-intensity NPPV of ≥6 hours

Exclusion Criteria:

1. Age <18 years
2. Excessive amount of respiratory secretions or weak cough
3. Upper airway obstruction
4. Recent oral, facial, or cranial trauma or surgery; recent gastric or esophageal surgery
5. Potential risk factors for restrictive ventilatory dysfunction (eg, consolidation or removal of at least one pulmonary lobe, massive pleural effusion, chest wall deformity, continuous strapping with thoracic or abdominal bandage, and severe abdominal distention)
6. Active upper gastrointestinal bleeding
7. Cardiac or respiratory arrest
8. Arterial oxygen tension/fraction of inspired oxygen <100 mmHg
9. Pneumothorax
10. Severe ventricular arrhythmia or myocardial ischemia
11. Severe hemodynamic instability despite fluid repletion and use of vasoactive agents
12. Severe metabolic acidosis
13. Refusal to receive NPPV
14. Endotracheal intubation already performed before ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
PaCO2 measured at 24 hours after enrollment | 24 hours
  PaCO2 measured at 24 hours after enrollment.

SECONDARY OUTCOMES:
PaCO2 measured at 2 hours after enrollment | 2 hours
  PaCO2 measured at 2 hours after enrollment
PaCO2 measured at 6 hours after enrollment | 6 hours
  PaCO2 measured at 6 hours after enrollment
PaCO2 measured at 48 hours after enrollment | 48 hours
  PaCO2 measured at 48 hours after enrollment
PaCO2 measured at 72 hours after enrollment | 72 hours
  PaCO2 measured at 72 hours after enrollment
Glasgow coma scale score | 72 hours
  The glasgow coma scale score, ranging from 3 (coma) to 15 (normal consciousness), will be used to assess the consciousness level.
ΔPes | 72 hours
  Inspiratory esophageal pressure swing
Dyspnea score | 72 hours
  The dyspnea score will be assessed using a verbal analogue scale with levels from 0 (no dyspnea) to 10 (maximum dyspnea).
NPPV tolerance score | 72 hours
  NPPV tolerance will be recorded on a 4-point scale and then dichotomized into acceptable (score of 2 or 3) or poor (score of 0 or 1) tolerance.
Plasma level of TNF-α | 72 hours
  Plasma level of TNF-α
Plasma level of I-1β | 72 hours
  Plasma level of IL-1β
Plasma level of IL-6 | 72 hours
  Plasma level of IL-6
Plasma level of IL-8 | 72 hours
  Plasma level of IL-8
Plasma level of IL-10 | 72 hours
  Plasma level of IL-10

CONTACTS AND LOCATIONS:
Overall Officials: Zujin Luo, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, China

REFERENCES:
- [Derived] Luo Z, Cao Z, Li Y, Jin J, Sun W, Zhu J, Zhao N, Liu J, Wei B, Hu Y, Zhang Y, Ma Y, Wang C. Physiological effects of high-intensity versus low-intensity noninvasive positive pressure ventilation in patients with acute exacerbation of chronic obstructive pulmonary disease: a randomised controlled trial. Ann Intensive Care. 2022 May 19;12(1):41. doi: 10.1186/s13613-022-01018-4. PMID 35587843